CLINICAL TRIAL: NCT02761616
Title: A Study to Determine Biopsy Rate in Participants With a First Relapse of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML30038
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- eBC treated participants: Participants with metastatic disease after previously being treated for eBC were observed for 24 months.
  Interventions: Other: eBC treated participants

INTERVENTIONS:
Other: eBC treated participants — No intervention administered in this retrospective observational study.

SUMMARY:
This is a retrospective, and observational cohort study to determine the proportion of breast cancer first relapses, that are biopsied. The duration of the study will be approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed breast cancer treated for early breast cancer (eBC) with first metastatic relapse disease in the period from January 1, 2014 and December 31, 2015

Exclusion Criteria:

Not Applicable

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a first relapse of breast cancer after being treated for eBC.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2016-06; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of biopsied participants with metastatic relapse | Approximately up to 24 months

SECONDARY OUTCOMES:
Percentage of non-biopsied participants at first relapse according to different reasons for not performing a biopsy of the metastasis | Approximately up to 24 months
Percentage of biopsied and non-biopsied participants at first relapse metastatic breast cancer (mBC) for each metastatic site | Approximately up to 24 months
Percentage of biopsied participants at first relapse mBC according to each biopsy method | Approximately up to 24 months
Percentage of biopsied and non- biopsied participants at first relapse mBC for each molecular profile of primary tumor | Approximately up to 24 months
Percentage of biopsied participants at first relapse mBC for each molecular profile of biopsied metastases | Approximately up to 24 months
Percentage of biopsied participants at first relapse mBC with same and different molecular profiles between primary tumor and metastasis for each molecular profile | Approximately up to 24 months
Time to relapse | Approximately up to 24 months
Percentage of participants with type of first line therapy selected for metastatic disease | Approximately up to 24 months
Percentage of participants influenced with biopsy in mBC | Approximately up to 24 months
Percentage of biopsied and non- biopsied participants at first relapse mBC for each systemic treatment scheme in the adjuvant and in the metastatic setting | Approximately up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Argentina (4):
  - Cemic; Oncologia Clinica, Buenos Aires
  - Hospital de Morón, Morón
  - CENICLAR, Rosario
  - Centro Medico San Roque, San Miguel de Tucumán